CLINICAL TRIAL: NCT04308460
Title: Prospective Randomized Study Between Arthrocentesis and Operative Arthroscopy in the Management of Temporomandibular Joint Internal Derangement
Brief Title: Arthrocentesis Versus Operative Arthroscopy Treatment of TMJ Internal Derangement (TMJ)
Acronym: TMJ
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hams Hamed Abdelrahman (Other)
Responsible Party: Sponsor-Investigator, Hams Hamed Abdelrahman, Assistant lecturer, Alexandria University
Organization: Alexandria University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: arthrocenetesis vs arthroscopy
Record Dates: First submitted 2020-03-08; First posted 2020-03-16 (Actual); Last update posted 2020-03-16 (Actual); Status verified 2020-03

CONDITIONS: Temporomandibular Joint Disc Displacement; Temporomandibular Joint Disorders
Keywords: TMJ, TMJ arthroscopy, arthroscopy, arthrocentesis
MeSH Terms: conditions — Temporomandibular Joint Disorders | interventions — Arthrocentesis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- arthrocentesis group (Active Comparator): the group of internal derangement patients which was treated with arthrocentesis procedure
  Interventions: Procedure: arthrocentesis
- operative arthroscopy group (Active Comparator): the group of internal derangement patients which was treated with operative arthroscopy procedure
  Interventions: Procedure: operative arthroscopy

INTERVENTIONS:
Procedure: arthrocentesis — lavage of the temporomandibular joint was done
  Arms: arthrocentesis group
Procedure: operative arthroscopy — operative intervention inside the temporomandibular joint was done using arthroscope
  Arms: operative arthroscopy group

SUMMARY:
Introduction: Temporomandibular disorders (TMDs) are relatively common conditions and internal derangement is the most common among them. Different methods have been suggested for treatment , beginning with conservative approaches ending with surgery. Nowadays, arthroscopy and arthrocentesis have eliminated the use of many of the more complex surgical procedures. Despite such advancements, there is lack of prospective, randomized, clinical studies to support the use of either both. In doing the necessary studies, and comparing the results, it will be important to develop standardized patient selection criteria and treatment options to be used by all investigators.

Objectives: To compare between arthrocentesis and operative arthroscopy in the management of patients with internal derangement of temporomandibular joint stage II and III Wilkes.

Materials and Methods: a prospective study was done on 40 patients with temporomandibular joint internal derangement and were divided into 2 groups, 20 patients were treated with arthrocentesis and 20 patients were treated with operative arthroscopy.

DETAILED DESCRIPTION:
The temporomandibular joint (TMJ) is known as ginglymo-arthrodial joint and is formed by the bony articulations of the mandibular condyle with the glenoid fossa of the temporal bone. Interposed between the condyle and the fossa is a piece of dense avascular fibrous connective tissue namely the TMJ disc which divides the joint into superior and inferior compartments.

TMJ disorders are relatively common conditions with incidence rate of 28% - 88%. They affect up to one-third of all adults at some stage in their life.

Two fundamental components form the temporomandibular system, the temporomandibular joint (TMJ) and the associated neuromuscular system. Any defect of one or both components lead to temporomandibular disorder (TMD). Symptoms can be unilateral or bilateral involving the face, head or jaw. TMDs are broadly divided by the American Academy of Orofacial Pain (AAOP) into muscle related TMD (myogenous), and joint-related TMD (arthrogenous). The two types can be present concurently, making diagnosis and treatment more testing.

Internal derangement of the temporomandibular joint (TMJ) is one of the most common temporomandibular disorders. It was defined by Dolwick in 1983 as an abnormal relation between the temporomandibular disc with respect to the temporal fossa, the mandibular condyle, and the temporal eminence of the TMJ. It may be present with anterior disc displacement, with or without reduction, perforation of the the articular disc or even the retrodiscal tissue, and degenerative changes of the joint surfaces. Clinically, it is usually accompanied by clicking, pain, limitation of mouth opening, and locking.

In 1989, Wilkes first established a classification which consists of 5 stages based on clinical, radiologic, and intraoperative findings.

Many methods have been suggested to treat this entity, beginning with conservative approaches. Medical treatment depending on nonsteroidal anti-inflammatory drugs (NSAIDs) and muscle relaxants, Occlusal splint therapy, and physical treatment are the most frequent options used among the conservative methods. Those refractory cases in which there was no effective improvement in terms of mandibular function and pain are amenable to further surgical treatment.

Initially, surgical treatment consisted of a discectomy, regardless of the type of internal derangement that was present . However, in 1979, Farrar and McCarty described surgical repositioning of the disc (discoplasty), showing that it was not necessary to remove the disc in most instances .

During the period when most surgeons were performing open surgical procedures for internal derangements of the TMJ, a small group of surgeons was beginning to experiment with arthroscopic surgery. First introduced by Ohnishi in 1975, this modality opened a new era in the diagnosis and treatment of such conditions.

Initially, arthroscopic treatment of patients with an internal derangement consisted mainly of lavage of the joint and later other intra-articular surgical manipulations such as lateral capsular release, and disc repositioning and fixation were added It has also become clear from the success of doing arthroscopic lysis of adhesions and lavage of the joint that disc position is less important than joint mobility and that patients can function successfully with an anteriorly displaced, non-reducing disc as a result of adaptation of the retrodiscal tissue and its acting as a pseudodisc It was an understanding of these two concepts that led to the introduction of arthrocentesis by Murakami and colleagues in l987 This technique was further refined by Nitzan et al., in 1991 Since that time, this procedure has largely supplanted arthroscopic lysis of adhesions and joint lavage as the initial approach to the management of majority of cases with internal derangements of the TMJ .

Nowadays, arthroscopy and arthrocentesis have eliminated the use of many of the more complex surgical procedures formerly used to manage intracapsular disease. Despite such advancements, however, clinicians are still encountering some difficulty in successfully treating many of these patients. review of the literature reveals that there is lack of prospective, randomized, clinical studies to support the use of either operative arthroscopy or arthrocentesis in the management of TMDs. In doing the necessary studies, and allowing for direct comparison of the results, it will be important to develop standardized patient selection criteria and treatment options to be used by all investigators .

The null hypothesis of the present study assumes that no significant difference will be found between operative arthroscopy and arthrocentesis in treating patients with Wilkes stage II and III internal derangement.

The aim of the study was to compare between arthrocentesis and operative arthroscopy in the management of patients with internal derangement of temporomandibular joint.

This study was conducted on 40 patients with temporomandibular joint internal derangement. Patients were admitted, investigated and managed in two departments:

1. Maxillofacial and Plastic Surgery Department, Faculty of Dentistry, Alexandria University, Egypt.
2. Oral and Maxillofacial Surgery Department, University Hospital Infanta Cristina, University of Extremadura, Badajoz, Spain.

The study compared between arthrocentesis and operative arthroscopy in the following points:

1. Mouth opening measuring the maximal interincisal opening in millimeters.
2. Lateral excursion movement.
3. Protrusive movement.
4. Pain score using visual analogue scale (VAS) .
5. Presence or absence of clicking.
6. Operative time. Patient selection: Randomized clinical trial

The patients were randomized using computer based random allocation technique into two groups:

1. Group I: Twenty patients were treated with Arthrocentesis
2. Group II: Twenty patients were treated with Operative Arthroscopy Research subjects Inclusion criteria The patients with TMJ internal derangement was divided into 5 stages according to Wilkes Classification. Only patients with stages II and III was included in this study.

Exclusion criteria

1. Medically unfit patients.
2. Stages I, IV & V Wilkes (Stage I patients will get benefit from conservative treatment and stage IV and V represent an advanced stages).
3. Patients with TMDs secondary to malocclusion.
4. Psychological instability.
5. Patients operated before for other TMJ problems. All patients were subjected to full history taking including medical and dental history, full clinical examination: general and TMJ examination, routine laboratory investigations and preoperative MRI.

Surgical technique A-Arthrocentesis

The procedure will be carried out under local anesthesia:

1. The patient is seated at a 45-degree angle with the head turned towards the non-affected side to allow an easy approach to the joint. After proper preparation of the target side, the external auditory meatus is blocked with cotton wool soaked in paraffin oil. A line is drawn on the skin from the middle of the tragus to the outer canthus of the eye. Entry points are marked along this cantho-tragal line. The first point corresponding to glenoid fossa is marked 10 mm from the midtragus and 2 mm below this horizontal line, The second point correspond to the articular eminence is marked 10 mm in front of the first point and 10 mm below the line.
2. Local anesthesia is applied, avoiding intra-articular injection to permit controlled sampling of synovial fluid. A 19-gauge needle connected to a 1 ml syringe filled with lactated Ringer's solution is inserted into the superior joint compartment at the posterior site. The solution is injected and immediately aspirated, and this procedure is repeated two more times in order to obtain sufficient fluid for diagnostic and research purposes.
3. Next, 2-3 ml of Marcaine 0.5% or lignocaine 2 % is injected to distend the upper joint space and anesthetize the adjacent tissues. Another 19-gauge needle is inserted into the distended compartment in the area of the articular eminence (anterior entrance site), enabling free flow of Ringer's solution through the superior compartment. With a syringe, the solution is either injected directly in to the joint or an infusion bag containing lactated Ringer's solution placed about 1 meter above the temporomandibular joint level, is then connected to one of the needles to allow free flow of about 200 ml of fluid through the joint. On termination of the procedure sodium hyaluronate is injected into the joint, then the needles are removed.

B-Arthroscopic technique

1. All procedures will be done under general anesthesia
2. Instrumentation In all procedures, 1.9 mm, zero-degree optical device, sleeves, sharp and blunt perforators, adhesion knives, an exploratory probe, and a bipolar electrode (Karl Storz Endoscopy, Tuttlingen, Germany)
3. The triple-channel arthroscopic technique of McCain et al is used After the first puncture of the fossa, a systematic diagnostic arthroscopy is carried out. A second puncture is carried out aiming at the anterior recess under direct arthroscopic visualization.
4. Anterior release Through the working cannula additional local anesthesia is injected to avoid pain and to decrease bleeding; it can also reduce the risk of masticatory muscle nerve injury. A Knife, coblation or laser probe are used to cut the anterior attachment of the disc and the neighboring part of the lateral pterygoid muscle. The incision line is located approximately 2-3 mm anterior to the anterior band of the disc and is carried out across the whole width from medial to lateral. The depth of the anterior release is no more than 2 mm to avoid breaking large blood vessels and damaging the masticatory muscle nerve in the anteromedial synovium. A sharp trocar is inserted to release the fibres further.
5. Disc reduction After the anterior release is completed, the obturator is positioned at the anterior margin of the disc and the disc is pushed backwards. The obturator slides along the surface of the disc and arrives in the posterolateral recess. The retrodiscal tissue is pushed down inferiorly and posteriorly.

Postoperative management Antibiotics and nonsteroidal anti-inflammatory drugs are routinely prescribed for 3 days. The softness of the postoperative diet should be decreased slowly. Exercises to improve mouth opening are explained to the patient and start 1 week after operation.

In patients with significant postoperative occlusal changes, a splint is recommended. It is designed to raise the bite and prevent contact between upper and lower incisors and canines. Due to the resulting distalization of the bite force, joint loading is reduced, which contributes to the joint's rehabilitation. The appliance should be left in place around the clock during the first ten postoperative days, then used at night for four additional weeks.(24)

The follow up of all patients was done accessing :

* Pain using VAS (Visual Analogue Scale).
* Clicking (improvement or persistence).
* Range of motion including: maximal interincisal opening, lateral excursion movement and Protrusive movement

ELIGIBILITY:
Inclusion Criteria:

* The patients with TMJ internal derangement will be divided into 5 stages according to Wilkes Classification. Only patients with stages II and III will be included in this study.

Exclusion Criteria:

1. Medically unfit patients.
2. Stages I, IV & V Wilkes (Stage I patients will get benefit from conservative treatment and stage IV and V represent an advanced stages).
3. Patients with TMDs secondary to malocclusion.
4. Psychological instability.
5. Patients operated before for other TMJ problems.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2017-01-10 (Actual); Primary Completion 2019-06-10 (Actual); Study Completion 2019-12-16 (Actual)

PRIMARY OUTCOMES:
mouth opening | 6 months
  mouth opening was measured using the maximum interincisal opening in millimeter

SECONDARY OUTCOMES:
post operative pain score | 6 months
  pain was measured using the visual analogue scale from 0 to 10 where 10 is the worst pain and zero indicates no pain
protrusive movement | 6 months
  was measured in millimeter
lateral excursion movement | 6 months
  was measured in millimeter

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed H Warda, PhD, Study Director — Alexandria University; Mohamed M Fata, PhD, Principal Investigator — Alexandria University; Ahmed M Medra, PhD, Principal Investigator — Alexandria University; Florencio G Monje, PhD, Principal Investigator — University Hospital of badajoz, Sapin; Aly M Atteya, MS, Principal Investigator — Alexandria University
Locations (2):
- Alexandria Faculty of Dentistry, Alexandria, Egypt
- University Hospital of Badajoz, Badajoz, Spain

IPD SHARING:
Plan to Share IPD: Yes
The investigators are planning to share the methods and the results of this study with all the investigators
Supporting Information: Study Protocol, SAP
Time Frame: starting 6 months after publication
Access Criteria: the sharing access can be through PubMed when the study is published or through direct contact through this email: aly_atteya@hotmail.com